CLINICAL TRIAL: NCT03730935
Title: Effects of Respiratory Muscle Endurance Training on Blood Pressure, Exercise Performance and Sleep Quality in Healthy Elderly
Brief Title: Respiratory Muscle Endurance Training in Healthy Elderly
Acronym: RETE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RETE_2018
Record Dates: First submitted 2018-10-31; First posted 2018-11-05 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Respiratory muscle endurance training (30 minutes of volitional hyperpnoea at a target ventilation of 60-70% of the individual maximal voluntary ventilation for 5 days per week for 4 weeks).
  Interventions: Device: Respiratory muscle endurance training
- Sham (Sham Comparator): Sham training will be performed 5 times a week for 4 weeks using a mock asthma inhaler filled with 5.5 mg lactose powder. Subjects will be instructed to inhale the powder according to inhaler instructions and to then perform one full inspiration to total lung capacity using custom-made, low resistance tubing, which elicits minimal resistance to breathing.
  Interventions: Device: Respiratory muscle endurance training

INTERVENTIONS:
Device: Respiratory muscle endurance training — Respiratory muscle endurance training performed over the duration of 4 weeks

SUMMARY:
Prevalence of hypertension in the elderly is high. Given that hypertension is the leading cause of cardiovascular disease worldwide, safe and efficacious treatment options for this condition are highly desired. Apart from medication, changes in lifestyle are recommended to lower blood pressure, such as an increase in physical exercise. However, whole-body exercise is not feasible for all. Mobility disabilities, for example, increase sharply with age and are already common in middle age. For this population, it is necessary to have alternative, non-invasive interventions with similar effects on blood pressure. One such intervention might be respiratory muscle endurance training (RMET), but the effects on blood pressure are currently unknown.

The primary aim of this project is therefore to investigate the effects of RMET over the course of several weeks on resting blood pressure in healthy elderly. The secondary aim of the project is to evaluate the effects of RMET on uphill exercise performance in healthy active elderly given that elderly experience structural and functional changes of the lungs potentially affecting exercise performance. Finally, since prevalence of subjective sleep complaints is also high in the elderly, the present study will also investigate the effects of RMET on sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Age: 55-80 years
* Active (according to World Health Organisation Criteria)
* Systolic blood pressure lower than 140 mmHg and diastolic blood pressure lower than 90 mmHg
* Non-smoking
* Body-Mass-Index (BMI): 18.5-29.9 kg·m-2
* Normal lung function

Exclusion Criteria:

* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Intake of blood pressure medication or history of hypertension
* Intake of medications affecting sleep or the performance of the respiratory, cardiovascular or neuromuscular system
* Acute illness or chronic conditions affecting sleep or the performance of the respiratory, cardiovascular or neuromuscular system

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Blood pressure | At baseline and after completion of the study (approximately one month)
  Change in systolic and diastolic blood pressures (in mmHg) between baseline and after one month of training.
  Measurements will be done in triplicate after at least 10 minutes of quiet lying on a stretcher

SECONDARY OUTCOMES:
Incremental test | At baseline and after completion of the study (approximately one month)
  Change in exercise performance assessed with an incremental test to exhaustion (maximal oxygen consumption in ml· min-1· kg-1). The test will be conducted on a motorised treadmill.
Endurance capacity test | At baseline and after completion of the study (approximately one month)
  Change in exercise performance assessed with an endurance capacity test (time to exhaustion, in minutes). The test will be conducted on a motorised treadmill.
Sleep efficiency | At baseline between visits 1-2 and after completion of the study (approximately one month) at visits 4-5
  Change in sleep efficiency assessed with an actigraph device measuring sleep efficiency (in %), . Measurements will be done during the nights between the two baseline visits and between the two post visits
Sleep onset latency | At baseline between visits 1-2 and after completion of the study (approximately one month) at visits 4-5
  Change in sleep onset latency assessed objectively with an actigraph device measuring sleep onset latency (in min). Measurements will be done during the nights between the two baseline visits and between the two post visits
Fragmentation index | At baseline between visits 1-2 and after completion of the study (approximately one month) at visits 4-5
  Change in fragmentation index assessed objectively with an actigraph device measuring fragmentation index (unitless). Measurements will be done during the nights between the two baseline visits and between the two post visits
Oxygen saturation during the night | At baseline between visits 1-2 and after completion of the study (approximately one month) at visits 4-5
  Change in oxygen saturation assessed objectively with a wrist-worn pulse oximeter measuring oxygen saturation (in %). Measurements will be done during the nights between the two baseline visits and between the two post visits
Heart rate during the night | At baseline between visits 1-2 and after completion of the study (approximately one month) at visits 4-5
  Change in heart rate assessed objectively with a wrist-worn pulse oximeter measuring heart rate (in 1·min-1). Measurements will be done during the nights between the two baseline visits and between the two post visits
Subjective sleep quality | At baseline between visits 1-2 and after completion of the study (approximately one month) at visits 4-5
  Change in subjective sleep quality (i.e. "How well did you sleep?" and "How recovered are you?") measured at home after each intervention with a visual analog scale (VAS). The two VAS consists each of a 10cm-horizontal line, with the left end of the lines representing low sleep quality ("slept very badly" and "not recovered at all", respectively) and the right end representing good sleep quality ("slept very well" and "completely recovered", respectively). Participants are asked to draw a vertical line in between the two ends on each of the two VAS.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Physiology Lab, Institute of Human Movement Sciences and Sport, ETH Zurich, Zurich, Canton of Zurich, Switzerland